CLINICAL TRIAL: NCT02106169
Title: Impact of the Therapeutic Education on the Quality of Life of the Child From 8 to 12 Years Old (and His Family) Suffering of Food Allergy IgE-mediated.
Brief Title: Impact of the Therapeutic Education on the Quality of Life of the Child Suffering of Food Allergy IgE-mediated
Acronym: EducAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Society of Allergology (Unknown); Stallergenes laboratories (Unknown); Picot-Lactalis laboratory (Unknown); ALK Industries (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-A01104-41
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: IgE Mediated Food Allergy
Keywords: Food allergy; Children and families; Therapeutic education; Quality of life
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic education group (Experimental): At first, all patients will be invited to participate in a study of troop having for objective to estimate their quality of life. Then, the doctors offer patients randomized to therapeutic education to have a therapeutic education before the 4th month.
  The sessions will be led by a multidisciplinary equip. Each child and his family will have a therapeutic session (2 times 2 hours).
  Interventions: Behavioral: Therapeutic education group
- Control group (No Intervention): At first, all patients will be invited to participate in a study of troop having for objective to estimate their quality of life. Then, the patients randomized in this group will have the habitual medical care.

INTERVENTIONS:
Behavioral: Therapeutic education group
  Arms: Therapeutic education group

SUMMARY:
The purpose of the study is to determine whether therapeutic education can improve the quality of life of the child from 8 to 12 years old suffering of food allergy.

This study also show us if therapeutic education has an effect on the quality of life of child's family.

DETAILED DESCRIPTION:
Food allergy affects 5 - 6% of children. The major risk is anaphylaxis by ingestion of the forbidden allergen. The child and his family have to learn to deal with this risk. Therapeutic education can help the children to take care of their allergy.

Food allergy limits the child socialisation, leads to anxiety/fear, and impairs health-related quality of life. In the day of today, there is no cure treatment. Also, improve the quality of life is one of the goals of the food allergy management.

The impact of therapeutic education on quality of life has never been studied. We intend to study the impact of therapeutic education on the quality of life of children from 8 to 12 years old with IgE mediated food allergy.

Our hypothesis is the quality of life can be improved by therapeutic education.

ELIGIBILITY:
Inclusion Criteria:

* IgE mediated food allergy
* Child from 8 to 12 years old (included)
* Family who can have an internet access
* Children which parents have received study's information
* Child who can have a medical examination before inclusion (art. L.1121-11 du CSP).
* Patients who have a medical insurance.

Exclusion Criteria:

* Non IgE mediated food allergy
* Child with chronic disease, except asthma and atopic dermatitis
* Patients who already had a therapeutic education for food allergy
* Patient already included in another study

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

PRIMARY OUTCOMES:
Child FAQLQ global score | month 12

SECONDARY OUTCOMES:
Child FAQLQ global score | month 4
Child FAQLQ global score | month 6
All cause which can be influence the quality of life, especially occurrence of anaphylactic reactions | month 12
Parent FAQLQ global score | month 4
Parent FAQLQ global score | month 6
Parent FAQLQ global score | month 12

CONTACTS AND LOCATIONS:
Overall Officials: Chantal KARILA, MD, PhD, Principal Investigator — Necker hospital
Locations (1):
- Necker hospital, Paris, France